CLINICAL TRIAL: NCT01299220
Title: Pilot Study of Acitretin for Treatment of Erlotinib-induced Skin Rash
Brief Title: Study of Acitretin to Treat Skin Rash Caused by Erlotinib (a Chemotherapy Drug)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to enroll subjects by sponsor deadline
Sponsor: University of Pittsburgh (Other)
Collaborators: OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO10020317
Record Dates: First submitted 2011-02-15; First posted 2011-02-18 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Skin Rash
Keywords: Erlotinib; Acitretin; Rash; Dermatology; Oncology
MeSH Terms: conditions — Exanthema; Neoplasms | interventions — Acitretin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Acitretin — Acitretin 10 mg by mouth daily
  Other Names: Soriatane

SUMMARY:
This study will look at if a low-dose regimen of acitretin is helpful in treating a skin rash caused by the chemotherapy drug, erlotinib.

DETAILED DESCRIPTION:
This is a pilot trial with an initial target sample of 32 evaluable subjects. The study will last up to 12 weeks per subject and up to 9 months for the entire study. Cancer patients beginning antineoplastic therapy with the EGFR inhibitor erlotinib will be enrolled in this trial. Patients beginning erlotinib therapy will simultaneously initiate a skin care regimen consisting of twice daily application of Eucerin,TM Aveeno,TM or CeraveTM moisturizing cream and daily application of SPF 15 or greater sunscreen.

Those patients who develop rash of CTCAE Grade 2 or higher will be referred to us by their primary oncologist. Upon onset of the cutaneous eruption, the oncologist will initiate therapy with doxycycline (100 mg twice daily; those allergic to doxycycline will instead receive cephalexin, 250 mg twice daily).

On evaluation by the Principal Investigator, patients with insufficient response to a two week course of doxycycline (continued CTCAE Grade 2 or higher rash) will begin therapy with low-dose acitretin (10 mg/day). Patients will continue to receive 10 mg/day acitretin and will be followed for 12 weeks, after which they will be treated off-study according to an individualized regimen agreed upon by the patient and treating oncologist.

Patients who continue to have unacceptable skin eruptions and who require off-study dose reduction or interruption of erlotinib despite acitretin treatment, as well as those patients who develop CTCAE Grade 3 or higher toxicity presumptively due to acitretin, will be considered non-responders for this study. These patients will be treated off-study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older at the time of study enrollment.
* Started routine clinical, palliative, or experimental (off-label) treatment with erlotinib for solid tumors and have developed Grade 2 or higher skin toxicity based on National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.02.
* Failed therapy with a two-week course of antibiotic (doxycycline 100 mg twice daily, or cephalexin 250 mg twice daily in patients allergic to doxycycline).
* Willing and able to provide verbal and written informed consent
* If reproductive potential, both males and females,must practice effective contraceptive measures throughout the study. Women of childbearing potential must provide a negative pregnancy test (serum or urine) within 14 days prior to enrollment.

Exclusion Criteria:

* Pregnant or breast-feeding females.
* Known or suspected sensitivity to study medication.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 3 or worse.
* Treatment with a non-approved or investigational drug (with the exception of erlotinib used in an experimental setting) within 30 days prior to Day 1 of study treatment.
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated)for treatment of either a psychiatric or physical (e.g., infectious) illness.
* Bilirubin greater than or equal to three times the upper limit of normal. Sexually active women of childbearing potential must use an effective method of birth

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-11; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Lesion Counts | Baseline
  Lesion counts of the identified area of worst involvement will be done in a 5x5 cm area. All subsequent measurements will be done in the same 5x5 cm area.
Lesion counts | Change from baseline at week 1
  Lesion counts in area of worst involvement in 5x5 cm area
Lesion counts | Change from baseline at week 2
  Lesion count is performed in the worst area of involvement in 5x5 cm area
Lesion counts | Change from baseline at week 4
  Lesion count in the area of worst involvement in 5x5 cm area
Lesion count | Change from baseline at week 8
  Lesion counts in area of worst involvement in 5x5 cm area
Lesion counts | Change from baseline at week 12
  Lesion count in area of worst involvement in 5x5 cm area

SECONDARY OUTCOMES:
Quality of Life assessment | Baseline
  Standardized quality of life (QOL) tool will be used to assess impact of symptoms on QOL.
Quality of Life | Change from baseline at week 1
  Standardized QOL forms will be used
Quality of Life | Change from baseline at week 2
  Standardized QOL form will be used
Quality of Life | Change from baseline at week 4
  Standard QOL form will be used
Quality of Life | Change from baseline at week 8
  Standard QOL form will be used
Quality of Life | Change from baseline at week 12
  Standard QOL form will be used

CONTACTS AND LOCATIONS:
Overall Officials: Larisa J Geskin, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States